CLINICAL TRIAL: NCT05029024
Title: The Effect of a Single Session of 30-Minute Mindful Breathing in Reducing Fatigue Among Patients With Haematological Cancer - A Randomised Controlled Trial
Brief Title: Single Session of 30-Minute Mindful Breathing in Reducing Fatigue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Malaysia Sarawak (Other)
Collaborators: University of Malaya (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 201971-7588
Record Dates: First submitted 2021-08-04; First posted 2021-08-31 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Fatigue; Hematologic Malignancy
Keywords: Haematological cancer; fatigue; mindful breathing; Edmonton Symptom Assessment System
MeSH Terms: conditions — Fatigue; Hematologic Neoplasms | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Parallel-group, non-blinded, randomised control trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Active Comparator): Patients allocated to the intervention group received standard care plus a guided 30-minute mindful breathing session which consisted of four breathing exercises done consecutively in one-to-one manner. The four exercises included identifying the in-and out-breath, following the entire length of the breath, bringing the mind back to the body and relaxing the whole body. Each exercise lasted 7.5 minutes. Guidance was given by one of the two research assistants, who were medical doctors. They were trained by one of the co-investigators, who was a palliative care physician, certified in mindfulness training.
  Interventions: Other: 30-minute mindful breathing
- Control group (Placebo Comparator): Patients in the control group received standard care alone.
  Interventions: Other: control group

INTERVENTIONS:
Other: 30-minute mindful breathing — The four exercises included identifying the in-and out-breath, following the entire length of the breath, bringing the mind back to the body and relaxing the whole body. Each exercise lasted 7.5 minutes.
  Arms: Intervention group
Other: control group — standard care alone
  Arms: Control group

SUMMARY:
Investigators conducted a parallel-group, non-blinded, randomised control trial at the haemato-oncology unit of University Malaya Medical Centre, from 1st October 2019 to 31st May 2020. Patients included were ≥ 18 years, had histopathological diagnosis of haematological cancer, and fatigue score of ≥ 4 based on the fatigue subscale of Edmonton Symptom Assessment System (ESAS). Patients allocated to the intervention group received standard care plus a guided 30-minute mindful breathing session, while those in control group received standard care. The study outcomes include fatigue severity according to the fatigue subscale of ESAS, visual analogue scale of 0 - 10, and Functional Assessment of Chronic Illness Therapy Fatigue Scale Version 4, at minute 0 and minute 30.

DETAILED DESCRIPTION:
Investigators conducted a parallel-group, non-blinded, randomised control trial at the haemato-oncology unit of University Malaya Medical Centre (UMMC), a tertiary university hospital with 1,617 beds in Kuala Lumpur, capital of Malaysia, from 1st October 2019 to 31st May 2020. Patients included were aged 18 years and above, had a histopathological diagnosis of haematological cancer according to World Health Organisation classification, and a fatigue score of ≥ 4 based on the fatigue subscale of Edmonton Symptom Assessment System (ESAS). Patients were excluded if had impaired conscious level, cognitive impairment or any psychiatric illness that would prevent patients from giving informed consent or participate fully in the study; active or past history of cancer of other system, or a haemoglobin level of < 8g/dl.

Procedure:

Patients with haematological cancer attending the haematology clinic or admitted to the haematology ward of UMMC were consecutively screened for eligibility. The demographic and clinical data of the eligible patients, which include age, gender, ethnicity, religion, occupation, education level, marital status, type of haematological cancer, current status of cancer, types of cancer treatment, duration of cancer, blood parameters and other co-morbidities were obtained from the hospital Electronic Medical Record System. Any missing information was obtained by face-to-face interview with patients or relatives.

Patients who satisfied the inclusion criteria and agreed to participate in the study were randomly assigned into 2 groups based on computer-generated random numbers, in blocks of 10, with a one-to-one allocation ratio. Allocation sequence was concealed with sealed envelopes to prevent selection bias. Patients allocated to the intervention group received standard care plus a guided 30-minute mindful breathing session which consisted of four breathing exercises done consecutively in one-to-one manner. The four exercises included identifying the in-and out-breath, following the entire length of the breath, bringing the mind back to the body and relaxing the whole body. Each exercise lasted 7.5 minutes. Guidance was given by one of the two research assistants, who were medical doctors. The research assistants were trained by one of the co-investigators, who was a palliative care physician, certified in mindfulness training.

The training included a brief introduction to the basic concepts of mindfulness, followed by a 30-minute mindful breathing session guided by the trainer. Guidance on delivering the intervention with attention to paralanguage (intonation, rate and rhythm of speech, pitch, articulation, use of silence, etc.) and body language (eye contact, facial expression, posture and bodily movement), followed by supervision of the actual delivery of the 30-minute mindful breathing session by each research assistant were performed. The instructions for the 30-minute mindful breathing are presented in Table 1. Patients in the control group received standard care alone. Patients were allowed to resume usual activities 30 minutes prior to further assessment. Regardless of whether in intervention or control group, patients recruited in out-patient clinic were in sitting position, while patients recruited in ward were in lying position during the study.

The study outcomes were assessed at minute 0 (before intervention - T0) and minute 30 (after intervention - T30). The outcomes at T0 and T30 include fatigue severity according to the fatigue subscale of ESAS, a unidimensional visual analogue scale (VAS) of 0 - 10, and the score of Functional Assessment of Chronic Illness Therapy (FACIT) Fatigue Scale Version 4, a multidimensional fatigue scale. At the end of the study, patients in the intervention group were asked about feedback, any harm, and asked if patients were satisfied and willing to practise 30-minute mindful breathing in daily life.

The ESAS is a valid and reliable tool to assess nine common symptoms experienced by cancer patients. The nine symptoms assessed include: pain, tiredness, nausea, depression, anxiety, drowsiness, loss of appetite, wellbeing and shortness of breath. An additional blank scale is given to assess each patient's 'other problems' as needed. The severity for each symptom upon assessment has a rating from 0 to 10 on a numerical scale; with 0 indicating absence of the symptom and 10 indicating the worst symptom severity. For this study, the tiredness subscale was chosen to assess participants' fatigue severity.

The FACIT Fatigue Scale is a 13-item multidimensional assessment tool to measure individual's fatigue level during their normal daily activities over the past 7 days.(32) It has high internal validity (Cronbach's alpha = 0.96) and high test-retest reliability (ICC = 0.95). Each participant's level of fatigue is rated on a five point Likert scale (0 = not at all fatigued to 4 = very much fatigued). The total FACIT-fatigue score ranges from 0 to 52, with a higher score reflecting more fatigue.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 years and above
* had a histopathological diagnosis of haematological cancer according to World Health Organisation classification
* a fatigue score of ≥ 4 based on the fatigue subscale of Edmonton Symptom Assessment System

Exclusion Criteria:

* impaired conscious level
* cognitive impairment or any psychiatric illness that would prevent patients from giving informed consent or participate fully in the study
* active or past history of cancer of other systems
* a haemoglobin level of < 8g/dl

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
Fatigue severity by Edmonton Symptom Assessment System | 30-minute
  Fatigue severity according to the tiredness subscale of Edmonton Symptom Assessment System. The scale range 0 (no tiredness) to 10 (worst possible tiredness). The higher the value indicates the more tiredness/fatigue.
Fatigue severity by unidimensional visual analogue scale | 30-minute
  Fatigue severity according to the unidimensional visual analogue scale. The analogue scale range 0 - 10, the higher indicates the worst fatigue.
Fatigue severity by Functional Assessment of Chronic Illness Therapy Fatigue Scale Version 4 | 30-minute
  Fatigue severity according to the the score of Functional Assessment of Chronic Illness Therapy Fatigue Scale Version 4. This Scale has 13 items, each item range from 0 (not at all) to 4 (very much). The total score range from 0 to 52, the higher indicates more fatigue.

SECONDARY OUTCOMES:
General feedback | 30-minute
  General feedback was asses by using simple questionnaires designed by investigators. Patients were asked open ended questions about general feedback of the intervention, if the intervention was harmful, if patients were satisfied and willing to practise 30-minute mindful breathing in daily life.

CONTACTS AND LOCATIONS:
Overall Officials: Seng-Beng Tan, MBBS, Study Chair — Consultant, University Malaya Medical Center
Locations (1):
- Diana-Leh-Ching Ng, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ng DL, Gan GG, Anuar NA, Tung YZ, Lai NZ, Tan YW, Said SNM, Madihie A, Chai CS, Tan SB. The effect of a single session of 30-min mindful breathing in reducing fatigue among patients with haematological cancer - a randomised controlled trial. BMC Palliat Care. 2021 Oct 15;20(1):160. doi: 10.1186/s12904-021-00855-7. PMID 34649555

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-07-02): https://cdn.clinicaltrials.gov/large-docs/24/NCT05029024/Prot_SAP_000.pdf
  • Informed Consent Form (2019-07-02): https://cdn.clinicaltrials.gov/large-docs/24/NCT05029024/ICF_001.pdf